CLINICAL TRIAL: NCT05293275
Title: Virtual Reality as Nonpharmacologic Pain Management Among Hospitalized Inpatients. A Randomized Control Trial of Virtual Reality vs Standard of Care
Brief Title: Virtual Reality Pain Study
Acronym: VR Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Mark B Powers, Research Center Director Trauma Research Consortium, Baylor Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 021-367
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Hospitalized Patients 18 Years of Age or Older With Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Virtual Reality Group (Active Comparator): patients will use the virtual reality device over two days
  Interventions: Device: EaseVRx Virtual Reality Headset
- Standard of care (No Intervention): patients will receive standard of care only

INTERVENTIONS:
Device: EaseVRx Virtual Reality Headset — Virtual reality device with 360 degree visualization of various scenery and interactive modules
  Arms: Virtual Reality Group

SUMMARY:
Investigating pain in hospitalized patients in two groups: virtual reality usage group vs standard of care

DETAILED DESCRIPTION:
Patients will be randomized to either the virtual reality group or the standard of care group. The virtual reality group will use the device over two days. Both groups will answer questionnaires regarding their pain and anxiety. Medical records will be used to look at pain medication usage in both groups.

ELIGIBILITY:
Inclusion Criteria:

* • patients at least 18 years of age,

  * reported pain in last 24 hours ≥ 3 on the Numerical Rating Scales (NRS),
  * patients undergoing surgery,
  * expected hospital length of stay of at least 48 hours,
  * English fluency,
  * willing to comply with study procedures.
  * Hx opioid use

Exclusion Criteria:

* • gross cognitive impairment that would interfere with the ability to consent or complete study procedures

  * current or prior diagnosis of epilepsy, seizure disorder, dementia, or migraines,
  * hypersensitivity to flashing light or motion,
  * history of motion sickness or cyber sickness,
  * medical condition predisposing to or current nausea, vomiting or dizziness,
  * stereoscopic vision or severe hearing impairment,
  * injury to eyes, face or neck that impedes comfortable use of virtual reality,
  * cancer related pain,
  * PHQ-9 screen indicating suicidal ideation, patients will be referred to appropriate clinical intervention (see suicide protocol)
  * currently pregnant,
  * current or recent completion of participation in any interventional pain study (with in past 2 months)
  * substance abuse (alcohol or illegal drugs): Alcohol- NIAAA definition of heavy drinking as more than 4 drinks on any day or more than 14 drinks per week for men, more than 3 drinks on any day or more than 7 drinks per week for women. Any illegal drugs including marijuana

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by Numerical Pain Rating Scale | 3-4 days
  level of pain will be assessed using the Numerical Pain Rating Scale. The scale is composed of 0 (no pain) to 10 (worst pain imaginable)

SECONDARY OUTCOMES:
Anxiety assessed with numerical scale | 3-4 days
  level of anxiety assessed with numerical scale composed of 0 (no anxiety) to 10 (anxiety out of control)
The PROMIS sleep disturbance questionnaire | 3-4 days
  disruption of sleep assessed using the PROMIS sleep disturbance questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mark Powers, PhD, Principal Investigator — Research Center Director Trauma Research Consortium
Locations (3):
- United States (3):
  - Baylor Institute for Rehabilitation, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Baylor Scott and White Hospital-Temple, Temple, Texas